CLINICAL TRIAL: NCT01588574
Title: Study for Determine the Safety and Efficacy of Clostridium Botulinum Toxin Type A in Subjects With Cervical Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-GPRT-CD01
Record Dates: First submitted 2012-04-24; First posted 2012-05-01 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2013-02

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BOTOX (registered trade mark) (Active Comparator)
  Interventions: Biological: BOTOX(Registered trade mark)
- MT10109 (Experimental)
  Interventions: Biological: MT10109

INTERVENTIONS:
Biological: MT10109 — Botulinum toxin type A
  Arms: MT10109
Biological: BOTOX(Registered trade mark) — Botulinum toxin type A
  Arms: BOTOX (registered trade mark)

SUMMARY:
The purpose of this study is to determine the Optimal dose for safety and efficacy in the treatment of cervical dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18~75
* Have no clinically significant medical condition
* Cervical dystonia

Exclusion Criteria:

* Pregnant or lactation
* Subjects who have been administered the following drugs within the previous 1 month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Brisbane, Australia